CLINICAL TRIAL: NCT02120612
Title: Increasing Patient Knowledge of the Signs of Opioid Overdose and Naloxone in a Suburban Treatment Program
Status: Completed | Type: Observational
Sponsor: Edward Hospital (Other)
Responsible Party: Sponsor
Organization: Edward-Elmhurst Health System (Other)
Other Study IDs: LOH32414
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Opioid Dependence; Opioid Use Disorder
Keywords: Opioid Dependence; Addiction; Naloxone; Naloxone Education; Opiate Overdose Knowledge Scale; OOKS
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Historical Control Group: Historical Control Group will be assessed for knowledge prior to the implementation of the educational program.
- Naloxone Education Intervention Group: Group to begin receiving the Naloxone Education Intervention on the signs of opioid overdose and appropriate use of naloxone.
  Interventions: Other: Naloxone Education Intervention

INTERVENTIONS:
Other: Naloxone Education Intervention — The Naloxone Education Intervention is a curriculum that has been adapted from New York State Department of Health's, "Opioid Overdose Prevention" program for non-medical responders.
  Groups: Naloxone Education Intervention Group

SUMMARY:
The purpose of this study is to determine the effect that an educational intervention has on patient knowledge of the signs of opioid overdose and appropriate use of naloxone in a suburban outpatient treatment program.

DETAILED DESCRIPTION:
The outpatient Addiction Services program at Linden Oaks will begin implementing an educational program on the signs of opioid overdose and naloxone for all patients who have a diagnosis of opiate dependence in the investigators suburban treatment program. Subjects will be recruited from that population and administered a new, empirically validated scale (i.e. the Opiate Overdose Knowledge Scale; OOKS) both pre- and post-intervention to measure the effect that the educational program has on patient knowledge.

Patients will also be surveyed (i.e. History Survey) about their experiences over the previous 12-months (e.g. exposure to opiate overdoses, access/use of naloxone) prior to treatment; and, this History Survey will then be re-administered by phone, 1-3 months after discharge. The aim is to measure whether education influences patient behavior. Finally, all subjects will be administered an empirically-validated measure to assess subject shame and guilt (i.e. Guilt and Shame Proneness Scale; GASP), and response patterns in their behavior, to evaluate whether shame and guilt predict behavior at follow-up. The investigators will compare to data (i.e. OOKS, GASP, and History Survey) from a historical control group prior to the implementation of the educational program - and, also at 1-3 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects who have been diagnosed with a DSM opioid use disorder by LOH staff.

Exclusion Criteria:

* Subjects who are deemed to have moderate to severe cognitive impairment - as assessed by standard psychiatric evaluation from Linden Oaks clinical staff - will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects who have been diagnosed with a DSM opioid use disorder enrolled in an outpatient treatment program for the substance use disorder.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Opiate Overdose Knowledge Scale (OOKS) | 0-3 months
  The Opiate Overdose Knowledge Scale (OOKS) is an empirically-validated scale that measures knowledge of: (1) the risks, warning signs, and life-saving steps to take regarding an opioid overdose; and, (2) the appropriate use of naloxone.

SECONDARY OUTCOMES:
History Survey | 0-3 months
  The History Survey assesses subjects' experiences over the previous 12-months (e.g. exposure to opiate overdoses, access/use of naloxone).
Guilt and Shame Proneness Scale (GASP) | 0-3 months
  The Guilt and Shame Proneness Scale (GASP) is an empirically-validated measure to assess subject shame and guilt and behavioral response patterns.

CONTACTS AND LOCATIONS:
Overall Officials: David C Lott, M.D., Principal Investigator — Linden Oaks Hospital
Locations (1):
- Linden Oaks, Naperville, Illinois, United States